CLINICAL TRIAL: NCT06406478
Title: Measuring the Effects of Potential Work Time Schedule Changes on Nurse Manager Health and Patient Outcomes
Brief Title: Work Time Schedule Changes for Nurse Managers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jian Li, MD, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: #23-001694
Record Dates: First submitted 2024-04-10; First posted 2024-05-09 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-05

CONDITIONS: Work-Related Condition

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by study site and race, and then randomized into either the control or intervention group. The allocation sequences will be generated by a research team member using a random number table assigning groups 1:1, with equal numbers of participants in each intervention and control group.
Masking Description: No masking will occur in this study, as the groups will be aware of which schedule they are working, and the researchers will be examining differences between intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will begin working only four days a week as a schedule change.
  Interventions: Behavioral: Schedule Change
- Control Group (Active Comparator): The control group will continue to work five days per week, receiving standard practice for the schedule policies at the participating study sites.
  Interventions: Behavioral: No Schedule Change

INTERVENTIONS:
Behavioral: Schedule Change — This 4-day workweek is defined by any 4 ten hour shifts between Sunday and Saturday. It will be up to the discretion of participants in the intervention group to coordinate which 4 days they work. The 4 days will most likely be weekdays, but some participants may work weekends. If participants do any work from home, they will clock in remotely to account for the time.
  Arms: Intervention Group
Behavioral: No Schedule Change — The control group will continue to work five days per week, receiving standard practice for the schedule policies at the participating study sites.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to explore how working a 4-day schedule impacts nurse manager wellbeing and job performance. The main questions it aims to answer are:

* Do those working 4-days have improved wellbeing with reduced levels of burnout and work/family conflict when compared to those in the control group?
* Do levels of sleep, heart rate variability, and physical activity significantly differ between those working the 4-day schedule change and those in the control group?
* Are nurse manager satisfaction, patient satisfaction, and patient quality outcomes different among those working the 4-day schedule change and those in the control group?

Researchers will compare those working the 4-day schedule change to those working the standard 5-day schedule to determine causality between the intervention and the outcomes.

Participants will:

* Complete an initial visit to learn about the study.
* Begin wearing an OURA ring, which will collect data on physical activity, sleep, and heart rate variability. They will need to download the Oura Ring app on their phone and log in weekly to sync data so that the researchers may access it.
* Complete the first survey on the online REDCap platform (baseline).
* Begin the work schedule that was assigned to them.
* Clock in and out of work each shift.
* Take the follow-up survey online (month 3).
* Take the final survey online (month 6).

DETAILED DESCRIPTION:
Researchers are looking to measure the effects of potential worktime schedule changes on a) nurse manager wellbeing (i.e., work/family conflict, burnout) and b) job performance (i.e., nurse manager satisfaction, patient satisfaction, and patient quality outcomes). Informed by the Conservation of Resources (COR) theory, it is hypothesized that working 4 days per week instead of 5 will improve nurse manager wellbeing with reduced burnout and work/family conflict.

Using a randomized control trial design, nurse managers working at UCLA Health will be purposively recruited for the study. All participants will begin by taking a baseline online survey at the initial visit. This survey will collect primary data on wellbeing by measuring work/family conflict and burnout using the scales: Work-Family and Family-Work Conflict Scale + Work-Life Balance scale and the Oldenburg Burnout Inventory. The survey will include demographic questions and qualitative questions to elicit responses from nurse managers on how they believe the schedule changes impacts their wellbeing and job performance, providing additional understanding of results from the quantitative part of the survey. All participants will wear a biotracker, called an Oura Ring, for the study duration, uploading their data weekly via an app. The Oura Ring will provide primary data on sleep, heart rate variability, physical activity of nurse managers, which is hypothesized to mediate the relationship between the schedule change and nurse manager wellbeing. Secondary data will be gathered from UCLA MedNet system, including nurse manager TimeClock information, and de-identified aggregate data on job performance (including nurse manager satisfaction, patient satisfaction, and patient quality outcomes) over the duration of the study.

Participants will be randomized either into the intervention group or the control group at the initial visit. Those in the intervention group will begin working only four days a week as a schedule change, and those in the control will continue working five days per week. All participants will be taught how to input their time clock information on the UCLA Health System for all working days. Follow-up surveys will be completed remotely, occurring at three months and six months. The participants will receive a reminder email to complete the survey. After six months when the final survey is completed, study participation will conclude. Fifty participants are anticipated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Registered nurse
* Currently employed as a full-time nurse manager
* Having a span of control greater than 40 Full Time Equivalent (FTE) Direct Reports
* Currently working at either Ronald Regan UCLA Medical Center or UCLA Medical Center Santa Monica
* In the acute care setting

Exclusion Criteria:

* Those working in ambulatory care settings
* Nurse leaders with less than 30 FTE's
* Working part time
* Working a schedule less than 5 days a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
work family conflict | 0, 3, and 6 months
  Work family conflict will be measured with the Work-Family and Family-Work Conflict Scale + Work-Life Balance scale with 11 items. Work-Family Conflict is determined with a mean of score of responses for items 1 through 5; higher scores reflect more work-family conflict. Family-Work Conflict is determined with the mean of score of responses for items 6 through 10; higher scores reflect more family-work conflict. Work-Life Balance: Item score.
Burnout | 0, 3, and 6 months
  Burnout will be measured with the Oldenburg Burnout Inventory with 16 items. Disengagement in burnout is the sum of items: 1, 3(Reverse), 6(Reverse), 7, 9(Reverse), 11(Reverse), 13, and 15. Exhaustion is the sum of items: 2(Reverse), 4(Reverse), 5, 8(Reverse), 10, 12(Reverse), 14, and 16. Full Burnout is the sum of the two scales: Disengagement and exhaustion.

SECONDARY OUTCOMES:
Hospital rate of Central Line-associated Bloodstream Infection (CLABSI) | 6 months
  This variable is secondary, de-identified aggregate data from the UCLA Tableau server, narrowed down to location, date, and unit, and is a measure of Patient Quality Outcomes.
Hospital rate of center-association urinary tract infections (CAUTI) | 6 months
  This variable is secondary, de-identified aggregate data from the UCLA Tableau server, narrowed down to location, date, and unit, and is a measure of Patient Quality Outcomes.
Hospital rate of falls | 6 months
  This variable is secondary, de-identified aggregate data from the UCLA Tableau server, narrowed down to location, date, and unit, and is a measure of Patient Quality Outcomes.
Hospital rate of hospital acquired pressure injuries | 6 months
  This variable is secondary, de-identified aggregate data from the UCLA Tableau server, narrowed down to location, date, and unit, and is a measure of Patient Quality Outcomes.
Nurse manager satisfaction as assessed by the National Database of Nursing Quality Indicators (NDNQI) | 6 months
  This variable is secondary, de-identified aggregate data from the Center for Nursing Excellence stored on UCLA Health Box. This is measured by the National Database of Nursing Quality Indicators (NDNQI). NDNQI is the leading nursing-sensitive quality indicators database that contains unit-level information about 600+ measures relevant to nursing performance, patient and workforce experience, and health outcomes. The data is derived from a combination of administrative documentation and medical records. All information reported to NDNQI is available for NDNQI users to review and benchmark performance against other participating NDNQI facilities, to better understand how these findings stack up against competitors-providing valuable insights.
Patient satisfaction as assessed by the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAPHS) | 6 months
  This variable is secondary, de-identified aggregate data from the UCLA Tableau server. This is measured by the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAPHS). Individual patient responses are utilized for each of the ten HCAHPS measures for all valid and complete surveys within a discharge quarter. These measures include six composite items, two global items, and two individual items. The composite measures are each comprised of two to three questions from the HCAHPS survey.
  Composite Measures
  1. Communication with Nurses (Q1, Q2, Q3)
  2. Communication with Doctors (Q5, Q6, Q7)
  3. Responsiveness of Hospital Staff (Q4, Q11)
  4. Pain Management (Q13, Q14)
  5. Communication about Medicine (Q16, Q17)
  6. Discharge Information (Q19, Q20) Individual Items
  1. Cleanliness of Hospital Environment (Q8) 2. Quietness of Hospital Environment (Q9) Global Items
  1. Overall Hospital Rating (Q21)
  2. Recommend the Hospital (Q22)
Average weekly working hours | 3 and 6 months
  Time clock information will provide data for average weekly working hours
Oura Ring sleep score | 3 and 6 months
  Data will be collected from the Oura Ring. When participants open the Oura Ring app on their phones, their data will be shared with the researchers, providing a 30 day and 60 day summary score of sleep quality and duration. The Sleep Score ranges from 0-100.
  85 or higher: sleep is optimal. 70-84: sleep is good. Under 70: sleep is off and there may be lifestyle changes needed to improve it
Oura Ring heart rate variability | 3 and 6 months
  Data will be collected from the Oura Ring. When participants open the Oura Ring app on their phones, their data will be shared with the researchers, providing a 30 day and 60 day summary score of heart rate variability.
Oura Ring physical activity score | 3 and 6 months
  Data will be collected from the Oura Ring. When participants open the Oura Ring app on their phones, their data will be shared with the researchers, providing a 30 day and 60 day summary score of physical activity.
  The Activity Score ranges from 0-100 and tells participants at a glance, how to adjust their activity-rest balance:
  85 or higher: balance is optimal. 70-84: balance is good. Under 70: balance seems off and there may be lifestyle changes needed to improve it.
Write in questions: nurse manager perceptions of their work schedules | 3 and 6 months
  Nurse manager will have the opportunity to write in how they perceive their work schedules impact their own health and family life, and the outcomes of their patients. These questions are researcher-developed, allowing participants to share additional qualitative data.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Health, Santa Monica, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No